CLINICAL TRIAL: NCT01545284
Title: Pilot Study on the Use of Acitretin for the Treatment of Severe Chronic Hand Dermatitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Innovaderm Research Inc. (Other)
Collaborators: Tribute Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Inno-6022
Record Dates: First submitted 2012-02-29; First posted 2012-03-06 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Chronic Hand Dermatitis
Keywords: chronic hand dermatitis; acitretin; PGA
MeSH Terms: interventions — Acitretin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Acitretin (Experimental): Patients will receive acitretin once daily for a maximum of 24 weeks. Patients who reach a Physician Global Assessment (PGA) of clear or almost clear at week 12 will end the study. Patients who do not reach a PGA of clear or almost clear at week 12 will continue treatment up to week 24. The starting dose will be 10mg/day and, if well tolerated, it will be increased in the first 4 weeks to a maximum of 30 mg/day.
  Interventions: Drug: Acitretin

INTERVENTIONS:
Drug: Acitretin — All patients will receive open-label single oral acitretin 10 mg capsule once daily as a starting dose. If well tolerated, the dose will be increased in the first 4 weeks to a maximum of 30mg/day. Patients will be instructed to take the treatment as a single oral dose with a meal.
  Other Names: Soriatane

SUMMARY:
This pilot, phase II, 24-week study will recruit a total of 10 patients and will evaluate the efficacy and safety of acitretin in patients with severe chronic hand dermatitis .

DETAILED DESCRIPTION:
Patients will receive acitretin once daily for a maximum of 24 weeks. Patients who reach a Physician Global Assessment (PGA) of clear or almost clear at week 12 will end the study. Patients who do not reach a PGA of clear or almost clear at week 12 will continue treatment up to week 24. The starting dose will be 10mg/day and, if well tolerated, will be increased in the first 4 weeks to a maximum of 30 mg/day.

ELIGIBILITY:
Inclusion Criteria:

* Men or post-menopausal or surgically sterile women, 18 years of age or older at time of consent
* Has stable chronic hand dermatitis for at least 6 months
* Has chronic hand dermatitis with a PGA of severe at Day 0
* Unless vasectomized for at least 6 months or clinically diagnosed infertile, if male patient has a female partner of childbearing potential, patient and patient's partner are willing to use effective contraceptive method for at least 30 days before screening and until 2 years after the study. Male patient should not father a child or donate sperm during the study and for 2 years after the last treatment.

Effective contraceptive methods are:

* Barrier methods such as condom, sponge or diaphragm combined with spermicide in foam, gel or cream
* Female partner: Hormonal contraception (oral, intramuscular, implant or transdermal) which include Depo-Provera, Evra and Nuvaring. Oral contraceptives must have been taken at a stable dose for at least 90 days before study start
* Female partner: Intrauterine device (IUD)

  * Female patient has a negative serum pregnancy test within 14 days of Day 0
  * Capable of giving informed consent and the consent must be obtained prior to any study related procedures.

Exclusion Criteria:

* Female of childbearing potential, pregnant or lactating
* Has any other skin disease that could impair his/her safety during the study or interfere with the evaluation of the results
* Has a known allergy to acitretin, other retinoids or vitamin A derivates, or to any component of the study product
* Has used acitretin within 24 weeks of Day 0
* Has used systemic retinoid (including alitretinoin) within 6 months of Day 0
* Has used tetracycline or other vitamin supplements containing vitamin A within 4 weeks of Day 0
* Has used methotrexate within 6 months of Day 0
* Has used systemic therapy (e.g. corticosteroids, immunosuppressants or phototherapy) within four weeks of Day 0. Inhaled corticosteroids for stable medical conditions are allowed
* Has used any topical treatment for had dermatitis (e.g. retinoids, corticosteroids, tacrolimus, pimecrolimus) on the hands within 14 days of Day 0. If patients are using topical treatments for dermatitis on other areas of the body, it must be applied with gloves.
* Has used investigational agent within 30 days prior to Day 0, or within 5 half-lives of the investigational agent prior to day 0 (whichever is longer)
* Has a history of alcoholism or drug abuse within 12 months prior to Day 0
* Is planning to donate blood within 2 years after the end of the study
* Clinically significant increase in hepatic enzymes, cholesterol or triglyceride at screening that would, in the opinion of the investigator, put patient at risk if he/she receives acitretin
* Diagnosis or symptoms of inflammatory bowel diseases at screening or baseline
* Has an unstable or serious medical condition as defined by the investigator or presence of any significant medical condition, including severe renal impairment, that might cause this study to be detrimental to the patient
* Diagnosis or symptoms of active depression, including depression currently under control with medication, at screening or baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-03; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who reach a Physician Global Assessment (PGA) of clear or almost clear at the end of therapy. | 12-24 weeks

SECONDARY OUTCOMES:
Proportion of patients who reach a partial response defined as a PGA of clear, almost clear or mild at the end of therapy | 12-24 weeks
Change from baseline in modified Total Lesion Symptom Score (mTLSS) at the end of therapy | 12-24 weeks
Mean time to response defined as the number of days between baseline and the time the patient reaches a PGA of clear or almost clear | 24 weeks
Mean Patient Global Assessment (PaGA) at the end of therapy | 12-24 weeks
Change from baseline in extent of disease at the end of therapy | 12-24 weeks
Type, severity and relationship of adverse events | 12-24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bissonnette, MD, FRCPC, Principal Investigator — Innovaderm Research Inc.; Jerry Tan, MD, FRCPC, Study Director — Windsor Clinical Research Inc
Locations (2):
- Canada (2):
  - Windsor Clinical Research Inc., Windsor, Ontario
  - Innovaderm Research Inc., Montreal, Quebec